CLINICAL TRIAL: NCT06947707
Title: Safety and Efficacy of Edoxaban and Rivaroxaban to Cerebral Venous Thrombosis in Chinese Patients: A Prospective Cohort Study
Brief Title: Safety and Efficacy of Edoxaban and Rivaroxaban to Cerebral Venous Thrombosis in Chinese Patients
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Meng Ran, Professor, Xuanwu Hospital, Beijing
Other Study IDs: RMeng2
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Venous Thrombosis; Anticoagulants and Thrombotic Disorders; Anticoagulation Treatment; Anticoagulant Therapy; Anticoagulant Drugs; NOACs; Anticoagulant Prophylaxis/Therapy; Anticoagulation With NOAC; Anticoagulation With Direct Oral Anticoagulants
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- edoxaban
- Rivaroxaban

SUMMARY:
The goal of this observational study is to learn the safety and efficacy of edoxaban and rivaroxaban in Chinese population with the age range from 18 to 80 years who take edoxaban or rivaroxaban to treat their cerebral venous thrombosis (CVT). The main question it aims to answer are:

* Do cerebral veins or venous sinuses recanalize during the treatment period of edoxaban and rivaroxaban?
* Do the bleeding events occur during the treatment period of edoxaban and rivaroxaban?

The main tasks participants will be asked to do:

* Participants will comply fully with the prescribed regimen and take the edoxaban or rivaroxaban as directed at the specified dosage.
* Participants will return to hospital for scheduled follow-up assessments at months 3, 6, 9, and 12 post-enrollment to undergo face-to-face visits with investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged from 18 to 80 years and no gender preference;
2. Diagnosis of CVT as confirmed on MRBTI/MRV or CT/CTV or DSA;
3. Acute or subacute CVT from onset to door within 4 weeks;
4. The treating clinician irrelevant to the study is of the opinion that the patient is appropriate for edoxaban or rivaroxaban;
5. Patient or legally authorized representative is able to give written informed consent.

Exclusion Criteria:

1. Patient refuse to take edoxaban or rivaroxaban to treat CVT;
2. Pregnancy or breastfeeding women at the time of enrollment, or women who plan to get pregnant during study;
3. Patient is anticipated to require invasive procedure (e.g. thrombectomy, hemicraniectomy) prior to initiation of oral anticoagulation;
4. CVT secondary to central nervous system infection or severe head trauma;
5. It is in the proliferative stage of malignant tumors currently or within 6 months of diagnosis;
6. Bleeding diathesis or other contraindication to anticoagulation;
7. Any concurrent medical condition requiring mandatory antiplatelet or anticoagulant use;
8. Concomitant use of strong CYP3A4 or P-gp inhibitors;
9. Impaired renal function (CrCl<30 mL/min using Cockcroft-Gault equation) or investigator anticipate the CrCl lower than 30 mL/min during study;
10. Impaired liver function (ALT or AST exceeds twice the normal upper limit) or diagnosed as acute hepatitis currently;
11. Patient is unable to swallow due to depressed level of consciousness or other reasons;
12. Patient has a severe or fatal comorbid illness with life expectancy less than 6 months;
13. Patient with severe hypertension (SBP≥180mmHg and/or DBP≥110mmHg);
14. Patient is known to be allergic to edoxaban or rivaroxaban.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected CVT visited Xuanwu Hospital, Capital Medical University are evaluated from clinical symptoms, laboratory tests and neuroimaging findings. Eligible patients are screened according to the inclusion and exclusion criteria, and patients treated with edoxaban enter into "Edoxaban" group and with rivaroxaban into "Rivaroxaban" group.
Sampling Method: Non-Probability Sample
Enrollment: 1486 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recanalization of cerebral veins or venous sinuses | 1 year
major bleeding events | 1 year
  1. Symptomatic intracranial bleeding A new symptomatic intracranial hemorrhage OR worsening existing intracranial hemorrhage with a ≥33% change in hematoma volume, AND either an NIHSS score increase of 4 or more points, or a change in level of consciousness as per NIHSS item 1a, AND the clinical change is thought to be attributable to the hemorrhage.
  2. Other major bleeding Bleeding in a critical area or organ, including intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a drop in hemoglobin by 20 g/L or more, leading to transfusion of 2 or more units of whole blood or red cells.

SECONDARY OUTCOMES:
Venous thrombosis or recurrence of CVT | 1 year
  Venous thrombosis (including deep vein thrombosis or pulmonary embolism or visceral vein thrombosis) or recurrence of CVT (including new-onset CVT or progression of previous CVT)
Death or clinically relevant non-major bleeding events | 1 year
  Death related to venous thrombosis events or from other causes. A clinically relevant non-major bleeding event is an acute or subacute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of: (a) a hospital admission for bleeding, or (b) a physician guided medical or surgical treatment for bleeding, or (c) a change in antithrombotic therapy (including interruption or discontinuation of study drug).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No